CLINICAL TRIAL: NCT00935558
Title: Evaluation of p53peptide-pulsed Dendritic Cells in Combination With an Aromatase Inhibitor as a Treatment for Patients With Breast Cancer With Disease Recurrence After Adjuvant or First Line Endocrine Therapy.
Brief Title: Dendritic Cell Based Therapy for Breast Cancer Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no patients enrolled
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, Prof, MD, PhD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA 0822
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: dendritic cell; cancer vaccine; breast cancer; aromatase inhibitor; Zadaxin
MeSH Terms: conditions — Breast Neoplasms | interventions — lentiviral minigene vaccine of COVID-19 coronavirus; Thymalfasin; Interleukin-2; aldesleukin; exemestane; Anastrozole; Aromatase Inhibitors; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aromatase inhibitor and DC vaccination (Experimental): the HLA-A2 positive patients will be treated with AI, DC vaccines, Zadaxin and IL-2
  Interventions: Biological: DC vaccine
- Aromatase inhibitor (Active Comparator): the HLA-A2 negative patients will receive AI only
  Interventions: Biological: DC vaccine; Drug: aromatase inhibitor

INTERVENTIONS:
Biological: DC vaccine — DC vaccination regime consist of primary 10 intradermal injections of 1-2 weeks interval. At the time of each vaccine 6 MIU/m² IL-2 will be administered sc. Zadaxin 1.6 mg is injected sc twice a week. and tablet Aromatase inhibitor is administered ; Exemestane 25 mg (tablet) is administered PO daily or Femar 2,5 mg (tablet) is administered PO daily or Arimidex 1 mg (tablet) is administered PO daily
  Other Names: dendritic cell vaccine; Thymosin 1 alpha, Zadaxin®, Sigma-Tau; Interleukin-2, Proleukin®, Chiron B.V.; Aromatase inhibitor:Exemestane, (Aromasin®), Pfizer; or Femar®,letrozol, Novartis Healthcare; or Arimidex®, anastrozol, AstraZeneca
Drug: aromatase inhibitor — Exemestane 25 mg (tablet) is administered PO daily or Femar 2,5 mg (tablet) is administered PO daily or Arimidex 1 mg (tablet) is administered PO daily
  Other Names: Aromasin®, exemestane, Pfizer; Femar®, letrozol, Novartis Healthcare; Arimidex, anastrozol, AstraZeneca
  Arms: Aromatase inhibitor

SUMMARY:
The primary aim of this study is to investigate time to progression in breast cancer patients vaccinated with autologous dendritic cells pulsed with peptides in combination with adjuvant aromatase inhibitor (AI), Thymosin 1 alpha and interleukin-2. The secondary aim is to investigate whether a measurable immune response can be induced, and to evaluate the clinical effect (objective response rate) of the vaccination regime.

DETAILED DESCRIPTION:
Only patients who have tumors > 5 % positive for p53 by IHC can be referred to this treatment. All patients will receive standard dosage of AI +/- p53-DC vaccination. Patients who express HLA-A2 will also receive DC vaccination. Patients that do not express HLA-A2 will receive only AI and be regarded as controls.

The vaccination regime consists of primary 10 intradermal injections of 1-2 weeks interval (q1w x 4 → q2w x 6) with p53 peptide-pulsed dendritic cells, followed by monthly injections until progression; proleukin and Zadaxin are used as vaccine adjuvants.

Defined procedures are employed for generation of autologous dendritic cells for clinical application in a classified laboratory. Unmobilized leukapheresis will be used for isolation of large-scale mononuclear cells, and dendritic cells will be generated from monocytes by cytokine stimulation and loaded with p53 peptides. Frozen preparations of dendritic cells will be prepared using automated cryopreservation.Each patient will receive a minimum of 5x10^6 dendritic cells per treatment supplemented with interleukin-2 6 MIU/m² sc per vaccine and 1.6 mg Thymosin 1 alpha sc x 2/week.

Toxicity including autoimmunity will be evaluated using the common Toxicity Criteria (CTC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological proven metastatic or locally advanced ER+/PGR+ breast cancer in progression after receiving 1. line endocrine therapy.
* Further inclusion criteria: p53+ tumour, PS≤1, postmenopausal. Age >18, PS ≤ 1 and acceptable CBC and blood chemistry results

Exclusion Criteria:

* Patients with a history of any other neoplastic disease less than 5 years ago (excepting treated carcinoma in situ of the cervix and basal/squamous carcinoma of the skin)
* Patients with metastatic disease in the central nervous system
* Patients with other significant illness including severe allergy, asthma, DM, angina pectoris or congestive heart failure
* Patients with acute or chronic infection including HIV, hepatitis og TB
* Patients who received antineoplastic therapy including chemotherapy, radiation, immunotherapy or other agents, less than 4 weeks before the beginning of the trial
* Patients who received corticosteroids or other immunosuppressive agents
* Patients with active autoimmune diseases such as lupus erythematosus, rheumatoid arthritis or thyroiditis
* Severe hypercalcemia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To determine time to progression | after 8 and 16 weeks

SECONDARY OUTCOMES:
To evaluate safety of DC vaccination in combination with AI, to evaluate clinical tumor response, to evaluate treatment induced immune response to p53 end to evaluate duration of tumor and immune responses | Weekly the first 4 weeks, thereafter biweekly for five months, thereafter monthly

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, prof MD, Study Director — Department of Oncology, Copenhagen University Hospital, Herlev, Herlev Ringvej 75, DK-2730 Herlev; Denmark
Locations (1):
- Department of Oncology, Copenhagen University Hospital, Herlev, Herlev, Denmark

REFERENCES:
- [Background] Svane IM, Pedersen AE, Johansen JS, Johnsen HE, Nielsen D, Kamby C, Ottesen S, Balslev E, Gaarsdal E, Nikolajsen K, Claesson MH. Vaccination with p53 peptide-pulsed dendritic cells is associated with disease stabilization in patients with p53 expressing advanced breast cancer; monitoring of serum YKL-40 and IL-6 as response biomarkers. Cancer Immunol Immunother. 2007 Sep;56(9):1485-99. doi: 10.1007/s00262-007-0293-4. Epub 2007 Feb 7. PMID 17285289
- [Background] Svane IM, Pedersen AE, Johnsen HE, Nielsen D, Kamby C, Gaarsdal E, Nikolajsen K, Buus S, Claesson MH. Vaccination with p53-peptide-pulsed dendritic cells, of patients with advanced breast cancer: report from a phase I study. Cancer Immunol Immunother. 2004 Jul;53(7):633-41. doi: 10.1007/s00262-003-0493-5. Epub 2004 Feb 25. PMID 14985857